CLINICAL TRIAL: NCT06687590
Title: POst-Market ClINical Follow-up STudy of the SerranatOR PTA Serration Balloon CathEter
Brief Title: Serranator POINT FORCE Registry
Acronym: POINT FORCE
Status: Recruiting | Type: Observational
Sponsor: Cagent Vascular LLC (Industry)
Collaborators: Peachtree BioResearch Solutions Inc. (Unknown); Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CSP-0696
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Artery Disease (PAD); Dysfunctional AV Fistula; Dysfunctional AV Graft
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects: The study population will consist of subjects with claudication or ischemic rest pain, with de novo or restenotic lesions in the iliac, femoral, iliofemoral, popliteal, infrapopliteal and pedal arteries, or dysfunctional native or synthetic arteriovenous dialysis fistulae.
  Interventions: Device: Peripheral balloon angioplasty

INTERVENTIONS:
Device: Peripheral balloon angioplasty — Serration balloon angioplasty of iliac, femoral, iliofemoral, popliteal, infrapopliteal and pedal arteries, or dysfunctional native or synthetic arteriovenous dialysis fistula

SUMMARY:
The objective of this registry is to collect observational data under local standard of care and evaluate safety and performance of the Serranator® in treatment of peripheral artery disease (PAD), or dysfunctional native or synthetic arteriovenous dialysis fistulae in a real-world scenario.

The data and conclusions derived from this study will be used to provide clinical evidence for the clinical evaluation process.

ELIGIBILITY:
Inclusion Criteria:

* Subjects intended to be treated with Serranator® for de-novo or restenotic lesions of the iliac, femoral, iliofemoral, popliteal, infrapopliteal and pedal arteries or dysfunctional native or synthetic arteriovenous dialysis fistulae.
* Subjects presenting with claudication or critical limb-threatening ischemia (CLTI) by Rutherford Clinical Category 3, 4, 5, or 6 of the target limb.
* Age of subject is > 18.
* Subject or subject's legal representative has been informed of the nature of the study, agrees to participate and has signed the approved consent form.

Exclusion Criteria:

* Subjects with any medical condition that would make him/her an inappropriate candidate for treatment with Serranator® as per Instructions for Use (IFU) or investigator's opinion.
* Subject already enrolled in other investigational (interventional) studies that would interfere with study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects with claudication or ischemic rest pain, with de novo or restenotic lesions in the iliac, femoral, iliofemoral, popliteal, infrapopliteal and pedal arteries, or dysfunctional native or synthetic arteriovenous dialysis fistulae.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance Endpoint | Peri-procedural
  Device Success defined as the achievement of successful delivery, balloon inflation and deflation, and retrieval of the study device(s) with a post- Serranator® residual stenosis of ≤30% by angiographic core laboratory assessment at the intended target lesion.

SECONDARY OUTCOMES:
Safety Endpoint | Peri-procedural
  Major Adverse Events (MAE) until discharge, defined as all amputations and any re-intervention (surgical or endovascular) in the target limb.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States